CLINICAL TRIAL: NCT03738371
Title: Optimization of Performances During Thrombectomy Through In Situ Simulation
Brief Title: Formation of Health Professionals Through in Situ Simulation to Improve Performances During the Initial Step of Thrombectomy for Ischemic Strokes
Acronym: OPTISS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: OPTISS
Record Dates: First submitted 2018-09-28; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Time; Benefit of in Situ Simulation for This Kind of Training; Installation of the Patient Until the Percutaneous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Team of health professionals: Team of health professionals involved in thrombectomy (including specialized nurses in anesthesiology, anesthesiologists, neuroradiologist and technicians specialized in electro-radiology) will participate to in situ simulation.
  Interventions: Other: In situ simulation

INTERVENTIONS:
Other: In situ simulation — Team involved in thrombectomy procedures will be trained by in situ simulation. Simulation will reproduce the initial step of a thrombectomy procedure, i.e from from the installation of the patient to the percutaneous punch by the neuroradiologist. Simulation will be followed by a debriefing focused on the team performance. Three in situ simulation sessions will be realized by each team.

SUMMARY:
The thrombectomy is an emergency care provided as soon as possible to selected patients suffering from ischemic strokes. Many steps are necessary to prepare this specialized procedure of interventional neuroradiology, including installation and preparation of the patient for this act. This first and essential time required the intervention of many health professionals.

The approach consists of a series of formation through in situ simulations for these health professionals, in order to improve and optimize this first step of the procedure (from the installation of the patient to the percutaneous punch by the neuroradiologist).

ELIGIBILITY:
Inclusion Criteria:

* voluntary professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: health professionals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the team | 12 months
  Performance of the team will be scored using a technical and non-technical skill.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BAPTESTE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital neurologique, Centre Hospitalier Universitaire, Lyon, France